CLINICAL TRIAL: NCT03775889
Title: Engaging School and Family in Navajo Gardening for Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1001447; 8452 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dietary Habits; Eating Behavior; Health Behavior
MeSH Terms: conditions — Feeding Behavior; Health Behavior | interventions — Gardening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral (Experimental): Behavioral Gardening Exposure
  Interventions: Behavioral: Gardening

INTERVENTIONS:
Behavioral: Gardening — Assist with planting and maintaining the school garden, as well as observe the school garden curriculum and dietary assessment protocols

SUMMARY:
This study builds on several years of working with Navajo communities to increase gardening and healthy eating. In collaboration with the Dream Diné Charter School in Shiprock, NM, the investigators propose to develop a school garden intervention to increase fruit and vegetable consumption and reduce risk for obesity among Navajo families. The intervention will integrate: an enhanced school garden plot; a curriculum for elementary school children on gardening and healthy eating; and family engagement in the curriculum and at community gardening fairs.

ELIGIBILITY:
Inclusion Criteria:

* Attending School Participating in Trial
* Parent able to Participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Child healthy eating behaviors assessment | 1 year
  Assess servings of vegetables and fruits eaten per week from the picture sort frequency method using the 5 a Day questions

SECONDARY OUTCOMES:
Child Gardening Participation Survey | 1 year
  Survey children to see if they have a garden at home, and if so how often they do gardening activities there
Child Gardening Self-efficacy Survey | 1 year
  Survey children to identify how confident they are in their abilities to perform gardening behaviors, utilizing six-item likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Beresford, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No